CLINICAL TRIAL: NCT03697382
Title: Effect of Daily Ambulatory Activity on the Responses to Acute Aerobic Exercise.
Brief Title: Effect of Daily Steps on Fat Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Edward F. Coyle, Professor, University of Texas at Austin
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2018-08-0031
Record Dates: First submitted 2018-09-25; First posted 2018-10-05 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Atherosclerosis; Metabolic Syndrome
MeSH Terms: conditions — Atherosclerosis; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: Subjects will complete three experimental conditions which include 2 days of reduced step count (2,500, 5,000, and 7,500 steps/day) with 1-hour of exercise at 65% VO2max.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Very Low Steps (Experimental): Subjects will be asked to undergo reduced daily stepping to a level of 2,500 steps/d for 2 days. On the evening of day 2, they will be asked to run at 65% of VO2max for 1-hour.
  Interventions: Behavioral: Very Low Steps
- Low Steps (Experimental): Subjects will be asked to undergo reduced daily stepping to a level of 5,000 steps/d for 2 days. On the evening of day 2, they will be asked to run at 65% of VO2max for 1-hour.
  Interventions: Behavioral: Low Steps
- Moderate Steps (Experimental): Subjects will be asked to undergo reduced daily stepping to a level of 7,500 steps/d for 2 days. On the evening of day 2, they will be asked to run at 65% of VO2max for 1-hour.
  Interventions: Behavioral: Moderate Steps

INTERVENTIONS:
Behavioral: Very Low Steps — Subjects will have a 2-day control period during which step count and diet will be controlled for and recreated for the other trials. Following this 2-day period, they will undergo the Very Low Stepping trial with the acute bout of exercise on day 2. Day 3 will consist of the lipid tolerance test to determine the ability of the body to clear triglycerides.
  Arms: Very Low Steps
Behavioral: Low Steps — Subjects will have a 2-day control period during which step count and diet will be controlled for and recreated for the other trials. Following this 2-day period, they will undergo the Low Stepping trial with the acute bout of exercise on day 2. Day 3 will consist of the lipid tolerance test to determine the ability of the body to clear triglycerides.
  Arms: Low Steps
Behavioral: Moderate Steps — Subjects will have a 2-day control period during which step count and diet will be controlled for and recreated for the other trials. Following this 2-day period, they will undergo the Moderate Stepping trial with the acute bout of exercise on day 2. Day 3 will consist of the lipid tolerance test to determine the ability of the body to clear triglycerides.
  Arms: Moderate Steps

SUMMARY:
Reduced ambulatory activity has been shown to effect the response to a high fat tolerance test (HFTT) after acute exercise. This study will evaluate the effect of varying levels of daily ambulation on response to a HFTT after an acute aerobic exercise bout.

ELIGIBILITY:
Exclusion Criteria:

* Cardiovascular problems (e.g. pre-existing heart issues, coronary artery disease, hypertension, etc.)
* Respiratory problems
* Musculoskeletal problems that prevent prolonged sitting or exercise
* Obesity
* Susceptibility to fainting
* Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-09-29 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
6-Hour Plasma Triglyceride Area Under the Curve | 6-hours
  Areas under the curve for triglyceride concentration will be calculated for hourly samples from a 6-hour lipid tolerance test.

SECONDARY OUTCOMES:
6-Hour Plasma Insulin Area Under the Curve | 6-hours
  Areas under the curve for insulin concentration will be calculated for hourly samples from a 6-hour lipid tolerance test
6-Hour Plasma Glucose Area Under the Curve | 6-hours
  Areas under the curve for glucose concentration will be calculated for hourly samples from a 6-hour lipid tolerance test.

CONTACTS AND LOCATIONS:
Overall Officials: Heath Burton, M.S., Principal Investigator — University of Texas at Austin; Edward F Coyle, Ph.D., Study Director — University of Texas at Austin
Locations (1):
- University of Texas at Austin Human Performance Laboratory, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Burton HM, Coyle EF. Daily Step Count and Postprandial Fat Metabolism. Med Sci Sports Exerc. 2021 Feb 1;53(2):333-340. doi: 10.1249/MSS.0000000000002486. PMID 33105387